CLINICAL TRIAL: NCT03965676
Title: Evolution of Tophus and Erosions of Hands and Feet With Urate-lowering Therapy: Prospective Study Using Dual-Energy Computed Tomography
Brief Title: Evolution of Tophus and Erosions of Hands and Feet at DECT
Acronym: TOPHERO-CT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Canon U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180451
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-04

CONDITIONS: Tophaceous Gout
Keywords: Gout,Dual-energy computed tomography,Tophus,Erosion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult patients with a tophaceous gout (Other): Adult patients with a tophaceous gout but no urate-lowering treatment or treatment but target not reached (target = uricemia < 360µmol/L).
  Interventions: Other: Dual-Energy Computed Tomography examination

INTERVENTIONS:
Other: Dual-Energy Computed Tomography examination — Dual-Energy Computed Tomography examination at 6 and 12 months +/- 1 month of medical treatment with uricemia < 360μmol/L (baseline DECT is in the domain of usual care).

SUMMARY:
The main objective is to evaluate the decrease in crystalline volume of the target tophus using Dual-Energy Computed Tomography (DECT), after 6 months +/- 1 month of urate-lowering therapy with target uricemia.

Study hypothesis

* The dynamics of tophus resolution with urate-lowering therapy is poorly understood.
* It is variable according to the location of the tophus, peri articular / intratendinous, but also probably at the feet / hands, the initial overall volume of the tophus, the initial crystal charge of the tophus. Knowledge of prognostic factors for tophus resolution will help determine the best target for treatment follow-up for each patient.
* Erosions are the consequence of tophus. Tophus resolution could be associated with repair of erosions and stabilization of joint destruction.

DETAILED DESCRIPTION:
Study design The research is a non-randomized prospective bi-centric study in adult patients with tophaceous gout. It aims at studying tophus resolution (main objective), and prognostic factors for tophus resolution (secondary objective), and bone erosions, with Dual-Energy Computed Tomography (DECT) (secondary objective).

Study population

* Adult patients with a tophaceous gout but no urate-lowering treatment or treatment but target not reached (target = uricemia < 360µmol/L).
* Recruitment of patients during a visit or hospitalization in rheumatology at Lariboisière Hospital.

Calculated size of study population: 50 patients

No control group

Inclusion criteria

* Age greater than or equal to 18 years
* Patient with a tophaceous gout
* Without urate-lowering treatment or with treatment but uricemia not at target
* Having given its free and informed consent to participate in this study
* Affiliated with a social security system

Non-Inclusion criteria

* Pregnant or breastfeeding woman
* Participation in another intervention research or period of exclusion due to a previous research.
* Impossibility to position oneself in ventral position (position for hands/wrists DECT acquisition).

Acts or product added for the research study Dual-Energy Computed Tomography examination at 6 and 12 months +/- 1 month of medical treatment with uricemia < 360µmol/L (baseline DECT is in the domain of usual care).

For each patient, 3 visits (usual care):

* M0: Inclusion visit
* M6 + /- 1 month: visit, usual care, + DECT for research purpose
* M12 + /- 1 month: visit, usual care, + DECT for research purpose

Research duration:

* Inclusion period: 24 months
* Duration of participation (treatment + follow-up): 12 months + /- 1 month
* Total duration: 37 months

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Patient with a tophaceous gout
* Without urate-lowering treatment or with treatment but uricemia not at target
* Having given its free and informed consent to participate in this study
* Affiliated with a social security system

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Participation in another intervention research or period of exclusion due to a previous research.
* Impossibility to position oneself in ventral position (position for hands/wrists DECT acquisition).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-10-11 (Estimated)

PRIMARY OUTCOMES:
the percentage of decrease in crystal volume of the target tophus | after 6 months +/- 1 month of traitment
  decrease in crystal volume of the target tophus detected using dual-energy CT compared to the volume at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Richette Pascal, PhD, Principal Investigator — Rheumatology Department Lariboisière Hospital
Locations (2):
- France (2):
  - Radiology Department Lariboisière Hospital, Paris, Île-de-France Region
  - Reumatology Department Lariboisière Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No